CLINICAL TRIAL: NCT05282095
Title: Effect of HPV Integration on Prognosis of Young Women With CIN2 in China: A Multi-center Cohort Study in China
Brief Title: Effect of HPV Integration on Prognosis of Young Women With CIN2 in China
Status: Recruiting | Type: Observational
Sponsor: Fujian Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Binhua Dong, Principal Investigator, Fujian Maternity and Child Health Hospital
Other Study IDs: HPVZHCIN22021
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cervical Intraepithelial Neoplasia; HPV Infection; Virus Integration; HSIL, High Grade Squamous Intraepithelial Lesions
MeSH Terms: conditions — Uterine Cervical Dysplasia; Papillomavirus Infections; Squamous Intraepithelial Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples from cervix and vagina containing related cells, tissues and secretions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women aged from 18-45 with histopathologically confirmed CIN2: In the enrollment, women whose cervical histopathological results have been diagnosed as cervical intraepithelial neoplasia (CIN2) for the last 3 months with abnormal results will be included in this study. All participants will be followed up four, at 3th month, 6th month, 9th month and 12th month.
  Interventions: Other: Follow up

INTERVENTIONS:
Other: Follow up — Participants will be followed up at baseline, 3th, 6th, 9th and 12th months with HPV viral integration tests, HPV genotyping tests, thinprep cytologic tests (TCT) for cervix and vaginal secretion tests. Colposcopies and biopsies will be performed on the participants at 6 - and 12-month follow-up.

SUMMARY:
Clinically, cervical precancerous lesion is one of the important diseases that endanger the life safety and fertility of young women. Women with histopathologically confirmed CIN2 need regular HPV, cervical cytology, and colposcopic biopsy if necessary to assess the outcome and progression of the disease. In this study, we intend to visit Fujian Maternal and Child Health Hospital, Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology and other hospitals, including 300 CIN2 participants aged 45 and below diagnosed by histopathology, and collect the remaining cervical secretions and cervical exfoliated cell samples after clinical examination, even if you do not participate in this clinical study. In clinical diagnosis, treatment and follow-up, it is also necessary to collect the above specimens for relevant medical tests. Therefore, it is of great clinical and scientific significance to explore the role of HPV integrated detection in predicting the prognosis of young women with CIN2.

DETAILED DESCRIPTION:
This study aims to:1) determine the correlation between HPV integration and natural outcome in young CIN2 women. 2) determine the prognostic value of different HPV integration status in young women with CIN2. 3) determine the relationship between the integration status of different HPV genes in young CIN2 women and the results of vaginal flora and cervical exfoliative cytology. A prospective cohort of 300 participants under 45 years of age with histopathologically confirmed CIN2 was recruited from multiple centers, and HPV integration status, HPV infection status, cervical cytology, and vaginal flora diversity sequencing were performed at enrollment, 3 months, 6 months, 9 months, and 12 months. The purpose of this study was to evaluate the effect of HPV integration status and flora changes on the outcome and progression of CIN2 women, and to evaluate the correlation between HPV integration status and cervical cytology results.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 years of age or older and 45 years of age or younger, with a desire to conceive;
* Diagnosed with HSIL (CIN2) or HSIL (CIN2-3) via cervical tissue biopsy within the past 3 months, and has not undergone cervical surgery, physical, or medication treatment;
* The lesion area under colposcopy is less than 50% of the total cervical area within the past 3 months;
* Plans for 12-month follow-up observation for CIN2, with no surgical, physical, or medication treatment if the disease does not progress;
* Understands and voluntarily agrees to participate in the 12-month follow-up of this study, and signs the informed consent form.

Exclusion Criteria:

* Cervical status at the time of enrollment as determined by colposcopy within the past three months is Type III transformation zone;
* Pregnant or lactating;
* History of malignant reproductive tract tumors;
* History of hysterectomy, cervical surgery, or pelvic radiation therapy;
* Physical therapy to the cervix within 24 months prior to enrollment;
* The subject has a severe immune system disease that is active;
* Long-term use of contraceptives within 12 months prior to enrollment;
* Vaginal medication or irrigation within 72 hours prior to sampling (can re-enroll for sampling 3 days after cessation);
* Sexual intercourse within 24 hours prior to sampling (can re-enroll for sampling 24 hours after cessation);
* Received treatment for genital tract infections, HPV, or other STD pathogens within the past month (can re-enroll one month after cessation of treatment);
* Used antibiotics or vaginal microecological improvement products within the past month (can re-enroll one month after cessation of use);

Max Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: ≤45 years old Chinese women with cervical histopathology for CIN2.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Cervical histopathology testing at baseline | Baseline
  Cervical histopathology was performed at baseline for all participants.
Cervical histopathology testing at 6-month follow-up | 6-month follow-up
  Cervical histopathology was performed at 6-month follow-up for all participants.
Cervical histopathology testing at 12-month follow-up | 12-month follow-up
  Cervical histopathology was performed at 12-month follow-up for all participants.
Human Papillomavirus (HPV) viral integration test at baseline | Baseline
  Human Papillomavirus (HPV) viral integration test was performed at baseline for all participants.
Human Papillomavirus (HPV) viral integration test at 6-month follow-up | 6-month follow-up
  Human Papillomavirus (HPV) viral integration test was performed at 6-month follow-up for all participants.
Human Papillomavirus (HPV) viral integration test at 12-month follow-up | 12-month follow-up
  Human Papillomavirus (HPV) viral integration test was performed at 12-month follow-up for all participants.
Cervical cytology testing at baseline | Baseline
  All participants were tested for cervical cytology at the time of baseline.
Cervical cytology testing at 3-month follow-up | 3-month follow-up
  All participants were tested for cervical cytology at 3-month follow-up.
Cervical cytology testing at 6-month follow-up | 6-month follow-up
  All participants were tested for cervical cytology at 6-month follow-up
Cervical cytology testing at 9-month follow-up | 9-month follow-up
  All participants were tested for cervical cytology at 9-month follow-up
Cervical cytology testing at 12-month follow-up | 12-month follow-up
  All participants were tested for cervical cytology at 12-month follow-up
16SrRNA sequencing of the vaginal secretions at baseline | Baseline
  All participants underwent vaginal secretion sequencing at baseline.
16SrRNA sequencing of the vaginal secretions at 3-month follow-up | 3-month follow-up
  All participants underwent vaginal secretion sequencing at 3-month follow-up.
16SrRNA sequencing of the vaginal secretions at 6-month follow-up | 6-month follow-up
  All participants underwent vaginal secretion sequencing at 6-month follow-up
16SrRNA sequencing of the vaginal secretions at 9-month follow-up | 9-month follow-up
  All participants underwent vaginal secretion sequencing at 9-month follow-up
16SrRNA sequencing of the vaginal secretions at 12-month follow-up | 12-month follow-up
  All participants underwent vaginal secretion sequencing at 12-month follow-up
Human Papillomavirus (HPV) genotyping tests at baseline | Baseline
  All participants underwent Human Papillomavirus (HPV) genotyping tests at baseline.
Human Papillomavirus (HPV) genotyping tests at 3-month follow-up | 3-month follow-up
  All participants underwent Human Papillomavirus (HPV) genotyping tests at 3-month follow-up.
Human Papillomavirus (HPV) genotyping tests at 9-month follow-up | 9-month follow-up
  All participants underwent Human Papillomavirus (HPV) genotyping tests at 9-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Pengming Sun, Study Chair — Fujian Maternal and Child Health Hospital
Locations (20):
- China (20):
  - Fujian Maternity and Child Health Hospital, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Longyan First Hospital, Longyan, Fujian
  - The Second Hospital of Longyan, Longyan, Fujian
  - Ningde Municipal Hospital of Ningde Normal University, Ningde, Fujian
  - The First Hospital of Putian City, Putian, Fujian
  - The Affiliated Hospital of Putian University, Putian, Fujian
  - Sanming Second Hospital, Sanming, Fujian
  - Zhangzhou affiliated Hospital of Fujian Medical University, Zhangzhou, Fujian
  - Gansu Provincial Maternal and Child Health Care Hospital, Lanzhou, Gansu
  - Shenzhen Maternity and Child HealthCare Hospital, Shenzhen, Guangdong
  - Guiyang maternal and child health care hospital, Guiyang, Guizhou
  - Hubei Maternal and Child Health Care Hospital, Wuhan, Hubei
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Jiangxi maternal and Child Health Hospital, Nanchang, Jiangxi
  - Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality
  - Northwest Women's and Children's Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang

REFERENCES:
- [Derived] Zhang Y, Zhang Y, Hu T, Pu X, Dong B, Tuo X, Zou H, Zhang W, Lyu Q, Huang W, Xue H, Xu S, Osafo KS, Ren Y, Lin W, Su J, Huang X, Sun P. Effect of HPV integration on prognosis of young women with CIN2 in China: protocol for a multicentre prospective cohort study. BMJ Open. 2025 Apr 28;15(4):e093863. doi: 10.1136/bmjopen-2024-093863. PMID 40295124